CLINICAL TRIAL: NCT03378466
Title: Heparin AnticoaguLation to Improve Outcomes in Septic Shock: The HALO International Phase II RCT
Brief Title: Heparin Anticoagulation in Septic Shock
Acronym: HALO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: infeasible to continue due-to inability to recruit during the COVID-19 pandemic and grants coming to an end.
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CancerCare Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCA2017
Record Dates: First submitted 2017-11-09; First posted 2017-12-19 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-01

CONDITIONS: Septic Shock; Vasodilatory Shock
MeSH Terms: conditions — Shock, Septic | interventions — Heparin; vinyltriethoxysilane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unfractionated Heparin (UFH) (Experimental): UFH initiated at 18 IU/kg/hr
  Interventions: Drug: Unfractionated heparin
- Venous thromboprophylaxis (VTE) (Other): as per local standard
  Interventions: Other: Venous thromboprophylaxis (VTE)

INTERVENTIONS:
Drug: Unfractionated heparin — UFH initiated at 18 IU/kg/hr, dosed according to total body weight and pragmatically adjusted according to local institutional policy to achieve an activated partial thromboplastin (aPTT) of 1.5 to 2.5 times that of the reference aPTT value or anti-Xa values targeted to local practice levels. Duration of study intervention will be a maximum of 5 days (120 hours) or until vasopressors have been discontinued for 24 continuous hours. All participants will then receive venous thromboprophylaxis according to local practice.
  Other Names: Heparin
  Arms: Unfractionated Heparin (UFH)
Other: Venous thromboprophylaxis (VTE) — May include subcutaneous heparin or dalteparin, sequential compression device or graduated compression stockings
  Arms: Venous thromboprophylaxis (VTE)

SUMMARY:
This study is a pragmatic open-label international randomized trial comparing therapeutic dose intravenous unfractionated heparin (UFH) to standard care venous thromboprophylaxis in patients diagnosed with septic shock.

DETAILED DESCRIPTION:
Background and significance: Sepsis and septic shock account for 10% of admissions to the intensive care unit and constitute the second most frequent cause of death among admitted patients. The mortality rate associated with septic shock ranges from 30% to 50% and death is often due to multiple organ dysfunction coupled with systemic inflammation. Given the pathobiological relationship between coagulation and inflammation in sepsis, treatment with anticoagulants has been investigated in this population. Multiple lines of evidence suggest that heparin, a widely available, inexpensive anticoagulant, may improve clinical outcomes in sepsis, but high quality evidence to guide practice is lacking.

Hypothesis: Intravenous (IV) unfractionated heparin (UFH) reduces mortality and morbidity when administered to patients with suspected septic shock.

Study Design: A pragmatic open-label international randomized trial comparing therapeutic dose intravenous unfractionated heparin (UFH) to standard care venous thromboprophylaxis in patients diagnosed with septic shock.

Setting: To increase the external validity/generalizability of the trial results, 20 sites in 4 countries will participate.

Study Population: Patients with systemic inflammation, vasopressor dependent shock, and signs of organ dysfunction.

Interventions: IV infusion of UFH at 18 IU/kg/hr, dosed according to total body weight and pragmatically adjusted according to usual care to achieve an activated partial thromboplastin time (aPTT) of 1.5-2.5x that of the reference aPTT value (approximately 59-99 seconds). Alternately, therapeutic anti-Xa values (ie. values typically targeted for the treatment of venous thromboembolism) can be targeted based on local practice. Duration of heparin infusion is for a maximum of 5 days (120 hours) or until death, ICU discharge or discontinuation of vasopressors. The dose of UFH has been informed by our observational study and meta-analysis that showed a benefit of UFH in patients receiving therapeutic doses.

Control group: Local standard care for venous thromboprophylaxis (i.e. not therapeutic) which may include SC LMWH, SC UFH, sequential compression devices or graduated compression stockings.

Outcomes: At the end of the HALO international phase II trial, an international DSMB will be presented with by-group efficacy (vasopressor-free days) data in the context of 90-day mortality, and safety (bleeding and transfusion). With these data the DSMB will suggest: a) terminating enrollment for futility (lack of efficacy) or harm, or b) continuing to the phase III trial along with a recommended sample size to detect a clinically relevant difference in 90-day mortality. Patients will be analyzed according to the treatment group to which they are allocated. By-group data will remain blinded to study investigators so that these patients may be included in the HALO international phase III RCT. Our analytic approach provides a rationale to either stop, or to justify further investment in a large international phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Refractory hypotension documented within 18 hours prior to enrolment that requires the institution and ongoing use of vasopressor agents, (phenylephrine, norepinephrine, vasopressin, epinephrine, midodrine or dopamine >5 mcg/kg/min) at the time of enrolment. Refractory hypotension is defined as a systolic blood pressure (SBP) less than 90 mm Hg, or a systolic blood pressure more than 30 mm Hg below baseline, or a mean arterial pressure (MAP) less than 65 mm Hg and receipt of ≥ 2 litres of intravenous fluid for the treatment of hypotension (≥ 1 litre if dialysis dependent end-stage renal disease or if the patient is felt to be in congestive heart failure).
* At least 1 other new organ dysfunction (in addition to refractory hypotension), defined by the following:

  1. Creatinine ≥1.5x the known baseline creatinine, or ≥ 26.5 µmol/L increase or <0.5 mL/kg of urine output for 6-12 hours according to the KDIGO [Kidney Disease improving Global Outcomes (KDiGO)] guideline definition of acute kidney injury.
  2. Need for invasive mechanical ventilation or a P/F ratio <250
  3. Platelets <100 x109/L, or a drop of 50 x109/L in the 3 days prior to enrolment
  4. Arterial pH < 7.30 or base deficit > 5 mmol/L in association with a lactate > 4.0 mmol/L

Exclusion Criteria:

* Other forms of shock including cardiogenic, hemorrhagic, hypovolemic, neurogenic, or obstructive shock.
* Clinical suspicion or confirmation of a viral hemorrhagic shock syndrome including, but not limited to, dengue fever
* Rapid clinical improvement; vasopressors likely to be discontinued in the next 6 hours
* Received vasopressor therapy for greater than 18 hours prior to enrolment
* Bleeding Risk:

  1. Clinical: Active bleeding; head trauma; intracranial surgery or stroke within 3 months; history of intracerebral arteriovenous malformation, cerebral aneurysm or mass lesions of the central nervous system; history of a bleeding diatheses; gastrointestinal bleeding within 6 weeks; presence of an epidural or spinal catheter; selected cases of recent surgery where IV therapeutic UFH is considered contraindicated
  2. Laboratory: Platelet count <50 x109/L, INR >2.0, or baseline aPTT >50 seconds prior to enrolment
* Known or suspected adverse reaction to UFH including heparin induced thrombocytopenia (HIT).
* Use of any of the following treatments: UFH to treat a thrombotic event within 12 hours before enrolment; LMWH at a higher dose than recommended for prophylactic use within 12 hours before the infusion; warfarin (if used within 7 days before study entry AND if the INR exceeds 2.0 at enrolment); thrombolytic therapy within 3 previous days; use of IIb/IIIa inhibitors within the previous 7 days.
* Need for therapeutic anticoagulation
* Terminal illness with a life expectancy of less than 3 months, or no commitment to aggressive care.
* Consent declined from patient or authorized 3rd party
* Physician refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Vasopressor-free days. | 30 days
  The goal of phase II trial is to provide the international Data Safety Monitoring Committee (DSMC) with a sensible estimate to justify continued enrollment in an adaptive (sample size) trial. Vasopressor use, reflecting cardiovascular collapse due to overwhelming systematic inflammation, is a key inclusion criterion for the trial and durable discontinuation of such drugs and meaningful clinical improvement. Vasopressor-free days has been recommended as a preferred clinical outcome in phase II trials in critical illness.

SECONDARY OUTCOMES:
Clinical Outcome #1 - ICU mortality | From date of randomization until the first documentation of death from any cause or ICU discharge date or 90 days, whichever came first
  Survival
Clinical Outcome #2 - Hospital mortality | From date of randomization to the first documentation of death from any cause or hospital discharge date or 90 days, whichever came first.
  Survival
Clinical Outcome #3 - 90-day mortality | Up to day 90
  Survival
Clinical Outcome # 4 - ∆SOFA score (Sequential Organ Failure Assessment) | Daily from randomization to ICU discharge or hospital discharge or time of death or to study day 9 if still in ICU or hospital.
  Organ failure assessment using the SOFA scoring tool
Clinical Outcome # 5 - Hospital-free days to day 90 | from hospital admission to hospital discharge or time of death to day 90
  Hospital admission duration in the context of survival
Clinical Outcome #6 - Renal replacement therapy-free days to day 28 | from start of renal replacement therapy to study day 28
  Renal replacement therapy duration in the context of survival
Safety Outcome #1 - Major Bleeding | Assessed daily to day 8
  Rates of major bleeding using a validated bleeding assessment tool
Safety Outcome #2 - Minor Bleeding | Assessed daily to day 8
  Rates of minor bleeding using a validated bleeding assessment tool
Safety Outcome #3 - Suspected HIT (Heparin induced thrombocytopenia) | Assessed daily to day 8
  Incidence of any laboratory testing for HIT including screening or confirmatory tests
Safety Outcome #4 - Confirmed HIT (Heparin induced thrombocytopenia) | Assessed daily to day 8
  Postive confirmatory HIT test (one of Serotonin release assay (SRA) or Heparin induced platelet aggregation (HIPA))
Rate of enrolment | Monthly starting at individual site initiation through to end of enrollment, estimated two years
  average number of patients enrolled per site per month

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Zarychanski, MD MSc, Principal Investigator — University of Manitoba; Anand Kumar, MD, Principal Investigator — University of Manitoba; Dean A Fergusson, PhD MHA, Principal Investigator — University of Ottawa
Locations (51):
- Froedtert Hospital, Milwaukee, Wisconsin, United States
- Brazil (29):
  - Hospital Sao Jose, Altamira
  - Hospital Novo Atibaia, Atibaia
  - Hospital de Amor (Barretos), Barretos
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte
  - Hospital Tacchini, Bento Gonçalves
  - Hospital de Brasília, Brasília
  - Hospital Ortopedico e Medicina Especializada ltda. - HOME, Brasília
  - Instituto de Cardiologia do Distrito Federal, Brasília
  - Hospital Maternidade São José, Colatina
  - Hospital Baía Sul, Florianópolis
  - Hospital Nereu Ramos, Florianópolis
  - Hospital de Amor Jales, Jales
  - Unimed Cariri Hospital, Juazeiro do Norte
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto, Ribeirão Preto
  - Hospital Bruno Born, Rio Grande
  - Hospital da Cidade, Salvador
  - Santa Casa de São João Del Rei, São João del Rei
  - Hospital AC Camargo, São Paulo
  - Hospital Beneficência Portuguesa, São Paulo
  - Hospital da Luz, São Paulo
  - Hospital das Clinicas da faculdade de Medicina de Universidade de São Paulo, São Paulo
  - Hospital e Maternidade Sao Vicente, São Paulo
  - Hospital Santa Paula, São Paulo
  - Hospital Sepaco, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual de São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP, São Paulo
  - Hospital Ana Nery, Taguatinga
- Canada (11):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver Island Health Authority, Victoria, British Columbia
  - St Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Niagara Health System - St Catharines Site, Saint Catherines, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec - Universite Laval, Québec, Quebec
  - Hopital de l'Enfant-Jesus, Québec
- Greece (2):
  - ATTIKON University Hospital, Athens
  - Korgialeneion Benakeion Hospital, Athens
- AMRI Hospital Kolkata, Kolkata, India
- Pakistan (4):
  - Dr Ruth K.M. PFAU Civil Hospital, Karachi
  - Shaheed Mohtarma Benazir Bhutto Trauma Center, Karachi
  - The Indus Hospital, Karachi
  - Mayo Hospital Lahore, Lahore
- Philippines (3):
  - The Asian Hospital, Manila
  - The Medical City, Manila
  - The Philippines General Hospital, Manila